CLINICAL TRIAL: NCT04018950
Title: Single Period, Open Label, Phase 1 Study to Determine the Excretion and Metabolism of 14C-ETX2514 Administered Intravenously in Healthy Male Subjects
Brief Title: Study to Determine the Excretion and Metabolism of 14C-ETX2514 Administered Intravenously in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS2514-2018-0002
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Acinetobacter Baumannii-calcoaceticus Complex Infections
Keywords: Acinetobacter baumannii-calcoaceticus; complex infections; ETX2514; excretion; metabolism
MeSH Terms: interventions — durlobactam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ETX2514 and 14C-ETX2514 (Experimental): Participants will receive a single intravenous infusion of 1 gram non-labeled ETX2514 and 1 microCurie (µCi) of 14C-ETX2514 in normal saline, administered as a 3-hour infusion.
  Interventions: Drug: ETX2514; Drug: 14C-ETX2514

INTERVENTIONS:
Drug: ETX2514 — intravenous infusion
Drug: 14C-ETX2514 — intravenous infusion

SUMMARY:
This study will be conducted to determine the routes and rates of excretion of radio label arising from 14C-ETX2514 and to characterize metabolites of ETX2514 arising from 14C-ETX2514 administered intravenously in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants, between 18 and 55 years of age (inclusive) at the time of Screening
* Body mass index (BMI) ≥ 18.0 kilograms per meters squared (kg/m^2) and ≤ 32.0 kg/m^2 at Screening and weight between 55.0 and 100.0 kg (both inclusive) at Screening and Day -1
* Able to understand and willing to sign the Informed Consent Form (ICF), and willing and able to comply with the study restrictions and investigative site rules for participants
* Judged to be in good health in the opinion of the Investigator on the basis of a medical evaluation (including a physical examination, medical history, electrocardiograms vital signs, and the results of biochemistry and hematology tests and urinalysis carried out at Screening, Day -1 and pre-dose on Day 1) that does not reveal any clinically significant abnormality, which evaluation will consider acceptable the presence of a stable condition (e.g., hypertension, hyperlipidemia, diabetes mellitus, hypothyroidism) that may be under medical control (i.e., adequate and stable treatment) having no clinical consequences of the condition that, in the judgment of the Investigator, would increase risk to the participant's health by participating in this study or would increase risk of not achieving the study objectives
* Participants with normal renal function as evidenced by creatinine clearance (CLcr) estimated by Cockcroft Gault formula
* Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to Screening.
* Male participants with female partners of childbearing potential may be enrolled if they are:

  1. documented to be surgically sterile (vasectomy); or
  2. using two adequate forms of highly effective contraception (together with the female partner), out of which one will be a physical barrier (i.e., condom combined with partner oral contraceptive, implant, injectable, or indwelling intrauterine device), for 90 days after the study drug administration
* Must agree not to donate sperm from the Screening period through 90 days after the last dose
* Has sufficiently good venous access in both arms to confidently enable intravenous administration of study drug in one arm and serial blood sampling from the other arm
* Content of 14C in one or both (at Investigator's discretion) of urine and blood (or plasma) samples obtained at Screening does not significantly exceed the general environmental background 14C level

Exclusion Criteria:

* History or presence of oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, psychiatric or other disease or condition that in the Investigator's judgment poses a significant risk to the safety of the volunteer or the achievement of study objectives
* Clinically significant abnormal medical history, abnormal findings on physical examination, vital signs, electrocardiograms, or laboratory tests at Screening, Day -1 or pre-dose on Day 1 that the Investigator judges may put at risk achieving the objectives of the trial or protecting the safety of the volunteer
* History of cancer judged not to be in full remission for at least 5 years (except basal cell skin cancer or squamous cell skin cancer with history of curative treatment and no recurrence for at least 1 year prior to screening), as judged by the Investigator
* Any acute illness including clinically significant infection within 30 days prior to Screening
* Acute illness within 14 days prior to study drug administration unless mild in severity and enrollment is approved by both Investigator and Sponsor's medical representative
* Presence of active infection requiring antibiotic treatment
* History of multiple and/or severe allergies to drugs or foods or a history of anaphylactic reaction
* Uncontrolled hyperuricemia (serum uric acid > upper limit of normal [ULN])
* Concomitant use of medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) or to compete for renal tubular secretion (e.g., probenecid) within 60 days prior to study drug administration
* Documented congenital or acquired long QT syndrome
* Corrected QT interval (QTc) using Fridericia correction (QTcF) at Screening, Day -1, or pre-dose (Day 1) > 450 milliseconds
* Family history of long QT syndrome or of unexplained sudden death in a first-degree relative under age 50
* Uncontrolled treated/untreated hypertension (defined as a mean of 3 repeated measurements with approximately 5 minutes of resting time between each measurement for systolic blood pressure [SBP] ≥ 140 millimeters of mercury (mmHg) and/or diastolic blood pressure [DBP] ≥ 100 mmHg
* Current presence of clinically significant hypotension (systolic blood pressure [SBP] < 90 mmHg and/or diastolic blood pressure [DBP] < 50 mmHg)
* Positive alcohol breath test or urine drug screen test at screening and/or Day -1
* Recent history of incomplete bladder emptying with voiding or of awaking more than once at night to void
* Usual habit of less than one or more than three bowel movements per day
* Positive testing for human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C
* History or presence of alcohol or drug abuse within the 2 years prior to Screening
* Excessive intake of alcohol, defined as an average daily intake of greater than three units, or an average weekly intake of greater than 21 units (one unit is equivalent to 1 can or bottle [12 ounces (oz)] of beer, or 1 measure [1.5 oz] of spirits, or 1 glass [5 oz] of wine) in the last 6 months prior to Screening
* Use of any prescription (including proton pump inhibitors [PPIs] and diuretics) or non-prescription drugs, including over-the-counter medication, health supplements, non-routine vitamins and herbal products such as St. John's Wort, within 2 weeks prior to study drug administration unless discussed and agreed with the Sponsor's medical representative in writing. Use of the following may be allowed within the 2 weeks prior to study drug administration:

  1. Topically applied medication (eye and/or nose drops/spray or creams/ointment/lotion applied to skin);
  2. Occasional use of metoclopramide or ibuprofen;
  3. Use of multivitamins, vitamin C (allowed up to 7 days prior to study drug administration), and acetaminophen (allowed up to 3 days prior to study drug administration).
* Use of caffeine or other xanthine containing products (coffee, black tea, green tea, decaffeinated coffee, decaffeinated tea, colas, kola, chocolate, cacao, guarana, guayusa, yerba mate), Seville oranges (sour/bitter or "marmalade"), grapefruit or grapefruit juice within 48 hours prior to study drug dosing
* History or evidence of difficulty with venous access or adverse symptoms in donating blood
* Participation in another investigational drug trial within 30 days prior to study drug administration (or 5 times the half-life of any drug used in the prior study, whichever is longer) or exposure to more than three new investigational agents within 12 months prior to study drug administration
* Exposure to radiation for therapeutic or diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton) within the last 12 months prior to dosing of the investigational drug, or an occupationally exposed worker
* Participation in another clinical trial in which a [14C]-labeled drug was administered within the year prior to Day -1
* Donation or loss of more than 450 milliliters blood during the 3 months before the start of Screening
* Unwilling to avoid strenuous or unaccustomed activity, sunbathing, or contact sports within 96 hours (4 days) prior to entry in the clinic research center
* History of seizures, head injury with loss of consciousness or meningitis
* History of bleeding disorders
* Surgery within the past 3 months prior to Screening determined by the investigator to be clinically relevant
* Participants who have any of the following abnormalities on laboratory values at Screening or on Day -1 including:

  1. White blood cell count < 3000/millimeters cubed (mm^3), hemoglobin < 11 grams per deciliter (g/dL);
  2. Absolute neutrophil count < 1200/mm^3, platelet count < 120,000/mm^3;
  3. Serum Alkaline phosphatase (AP) > 1.5x ULN;
  4. Serum transaminase (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) > ULN
* Any other reason, condition or prior therapy, which, in the opinion of the Principal Investigator, would make the participant unsuitable for this study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Cumulative urinary recovery of total radioactivity | -12-0 hours (pre-dose), and at 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after the initiation of the intravenous (IV) dose
Cumulative fecal recovery of total radioactivity | -12-0 hours (pre-dose), and at 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after the initiation of the IV dose
Mass balance as a sum of the percent of total radioactivity recovered in urine and feces | urine: -12-0 hours (pre-dose), and at 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after the IV dose; feces: -12-0 hours (pre-dose), and at 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after the IV dose
Metabolite profiles in plasma | pre-dose (-30 minutes) and at 1, 2 (± 2 minutes), 3 (just prior to shutting off infusion), 4, 6, 8, 10, 12 (± 5 minutes), 18, 24, 36, 48, 72, 96, 120, 144, and 168 hours (± 10 minutes) after the initiation of the IV dose or early termination
Metabolite profiles in urine samples | -12-0 hours (pre-dose) and over the following collection periods: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120,120-144, and 144-168 hours after the initiation of the IV dose
Metabolite profiles in fecal samples | -12-0 hours (pre-dose) and over the following collection periods: 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after the initiation of the IV dose

SECONDARY OUTCOMES:
Number of participants with any treatment-emergent adverse event | up to Day 8
Number of participants with any clinically significant clinical laboratory evaluation | up to Day 8
Number of participants with any clinically significant vital sign measurement | up to Day 8
Number of participants with any clinically significant electrocardiogram finding | up to Day 8
Number of participants with any clinically significant physical examination finding | up to Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Clinical Pharmacology Center, Baltimore, Maryland, United States